CLINICAL TRIAL: NCT06869330
Title: Implementation and Effectiveness of a Psychosocial Intervention Among Registered PLHIV at Pakistan Institute of Medical Sciences (PIMS) Islamabad Pakistan.
Brief Title: Implementation and Effectiveness of a Psychosocial Intervention Among Registered People Living With HIV(HIV Patients) at Pakistan Institute of Medical Sciences (PIMS) Islamabad Pakistan.
Acronym: PLHIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Dr Israr khan, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F-5-2/2024(ERRC)/PIMS
Record Dates: First submitted 2025-03-04; First posted 2025-03-11 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-03

CONDITIONS: HIV Positive
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- "Implementation and Effectiveness of a Psychosocial Intervention Among Registered PLHIV at PIMS Isla (Experimental)
  Interventions: Behavioral: psychosocial

INTERVENTIONS:
Behavioral: psychosocial — Measure changes in mental health indicators like depression, anxiety, and stress levels using validated scales (e.g. DASS 21).

SUMMARY:
"Implementation and Effectiveness of a Psychosocial Intervention Among Registered PLHIV at PIMS Islamabad Pakistan." The study aims to evaluate the impact of a structured psychosocial intervention on the mental health and well-being of people living with HIV (PLHIV) registered at PIMS.

Study Highlights:

1. Participants: Registered PLHIV receiving care at PIMS.
2. Data Tools: Standardized measures (e.g., DASS-21, WHO-5 Well-Being Index).
3. Design: Randomized Control Trial (RCT) with intervention and control groups, including pre- and post-intervention assessments.
4. Ethical Approval: Approved by Pakistan Institute of Medical Sciences Pakistan Islamabad's Ethical Review Board

DETAILED DESCRIPTION:
"Implementation and Effectiveness of a Psychosocial Intervention Among Registered PLHIV at PIMS Islamabad Pakistan" The study aims to evaluate the impact of a structured psychosocial intervention on the mental health and well-being of people living with HIV (PLHIV) registered at PIMS.

Study Highlights:

1. Participants: Registered PLHIV receiving care at PIMS.
2. Data Tools: Standardized measures (e.g., DASS-21, WHO-5 Well-Being Index).
3. Design: Randomized Control Trial (RCT) with intervention and control groups, including pre- and post-intervention assessments.
4. Ethical Approval: Approved by Pakistan Institute of Medical Sciences Pakistan Islamabad's Ethical Review Board

ELIGIBILITY:
Inclusion Criteria:•

1:PLHIV who are registered at HIV Treatment Centre at PIMS Islamabad.

* 2:PLHIV who are registered and visiting for regular follow up
* 3:Participants willing to provide written informed consent.(Acceptance or willing of participants)

Exclusion Criteria:

* 1:PLHIV who are registered, but with other co morbidities like TB, Hepatitis BC, Cardiac issues etc.
* 2:PLHIV who are registered and admitted due to severe any co morbidities.
* 3:PLHIV who are registered and are already involved in other studies
* 4:PLHIV who are registered and have history of receiving any psychosocial support or counseling before this study.
* 5:Participants not willing to provide written informed consent.(Refusal of participants).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Transgender
Enrollment: 128 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
"Implementation and Effectiveness of a Psychosocial Intervention Among Registered PLHIV at PIMS Islamabad Pakistan | From enrollment to the end of intervention at 6 months.
  Measure changes in mental health indicators like depression, anxiety, and stress levels using validated scale (Depression, Anxiety and Stress scale 21). Minimum value is 0 and Maximum value is 3.Higher scores means a worse outcome.
"Implementation and Effectiveness of a Psychosocial Intervention Among Registered PLHIV at PIMS Islamabad Pakistan | From enrollment to the end of intervention at 6 months.
  : Assess overall wellbeing using validated scale(WHO-5 Well-Being Index.).Minimum value is 0 and maximum value is 5.Higher scores means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shahzad Ali khan, phd, Study Director — Health Services Academy, Islamabad, Pakistan
Locations (1):
- Pakistan Institute of Medical Sciences Islamabad Pakistan, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No
PARTICIPANT DATA IS CONFIDENTIAL

REFERENCES:
- [Background] Arundell LL, Barnett P, Buckman JEJ, Saunders R, Pilling S. The effectiveness of adapted psychological interventions for people from ethnic minority groups: A systematic review and conceptual typology. Clin Psychol Rev. 2021 Aug;88:102063. doi: 10.1016/j.cpr.2021.102063. Epub 2021 Jul 7. PMID 34265501
- See also: Related Info — https://doi.org/10.1016/j.cpr.2021.102063